CLINICAL TRIAL: NCT03763097
Title: Sonographic Evaluation of the Single-incision Needleless (Contasure-needleless®) Mini-sling Placement to Predict Success
Status: Completed | Type: Observational
Sponsor: Bartin State Hospital (Other Government)
Responsible Party: Principal Investigator, Murat Yassa, Principal Investigator, Bartin State Hospital
Other Study IDs: Ba2018-4
Record Dates: First submitted 2018-11-24; First posted 2018-12-04 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Urinary Incontinence,Stress
Keywords: pelvic floor ultrasonography; transperineal ultrasound; introital ultrasound; mini-sling; needleless; Urinary Incontinence,Stress
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- participants: Patients who are scheduled for single-incision needleless (Contasure-needleless®) mini-sling for their stress urinary incontinence. They will be assessed by Pelvic floor ultrasound
  Interventions: Diagnostic Test: Pelvic floor ultrasound

INTERVENTIONS:
Diagnostic Test: Pelvic floor ultrasound — Pelvic floor ultrasound will include transperineal and introital ultrasound

SUMMARY:
Transperineal ultrasonography is gaining importance in preoperative and postoperative evaluation of the patient with urinary incontinence with allowing well detailed information about the anterior compartment.

There is little evidence that transperineal sonography can aid surgeons to predict the success or failure after mid-urethral slings.

We aimed to investigate the efficacy of sonography in mini-sling operations to predict the success or failure.

DETAILED DESCRIPTION:
Women who are scheduled for anti-incontinence operation due to their stress urinary incontinence will be pre- and postoperatively evaluated by transperineal and introital ultrasound.

Patients will be followed for at least 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically stress urinary incontinence
* Patients who claim that their condition severely impair their quality of life
* Patients who are failed on conservative management (life style changes and pelvic floor exercises)

Exclusion Criteria:

* Patients who have unregulated diabetes mellitus (they will be included after appropriate and sustainable blood glucose regulation)
* Patients who have neurological condition that may affect the incontinence
* Patients who have psychiatric disease that may affect the subjective evaluation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have stress urinary incontinence and who are scheduled for needleless mini-sling operation.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2019-04-21 (Actual); Study Completion 2019-04-21 (Actual)

PRIMARY OUTCOMES:
The correlation of failure with the sonographic features of the mesh | Evaluation at postoperative 1st and 4th weeks
  Patients will be accepted as failure if their stress test is positive Sonographic features of the mesh includes the shape of the mesh, the distance to the mid-urethra, the position related to the proximal urethra and the angle between the mesh arms on coronal axis

SECONDARY OUTCOMES:
Nocturia | Evaluation at postoperative 1st and 4th weeks and preoperatively
  The nocturia episodes will be evaluated by a "non-validated" Likert scale (between 0-3). Minimum and minimum scores are between 0 and 3. "0" will mean no episode of urinating during the sleep. "1" will mean one episode of nocturia. "2" will mean two episodes of nocturia. "3" will mean three or more episodes of nocturia. Higher values represent worse outcome.
Urge symptoms | Evaluation at postoperative 1st and 4th weeks and preoperatively
  Michigan Incontinence Severity Index (M-ISI) scale will be used to assess subjective outcome including urge symptoms. This scale has ten items, consisting of a total M-ISI domain (the sum of items 1-8) and a distinct Bother domain (the sum of items 9 and 10). The total M-ISI score consists of three subdomains (items 1-3 for stress urinary incontinence [SUI], items 4-6 for urge urinary incontinence [UUI], and items 7 and 8 for Pad usage [PU]. The responses for each item range from 0 to 4 on a Likert-type scale, with higher values representing greater symptoms and greater bother. Total domain and subdomain scores are obtained by simply adding the respective answers. The minimally important difference has been determined for the following domains/subdomains: total M-ISI (4 points), SUI (2 points), UUI (2 points), and PU (1 point).
Subjective success | Evaluation at postoperative 1st and 4th weeks
  Patient Global Improvement of Improvement will be used to assess the subjective success
POP-Q | Evaluation at postoperative 1st and 4th weeks and preoperatively
  POP-Q measurements will be assessed to measure the pelvic floor prolapse if exist
Anterior compartment mobility distances | Evaluation at postoperative 1st and 4th weeks and preoperatively
  On maximal Valsalva maneuver: Bladder neck descent (mm), pubourethral distance (mm), urethral thickness (mm, measured at proximal, mid and distal portions) and urethral length (mm)
Anterior compartment mobility angles | Evaluation at postoperative 1st and 4th weeks and preoperatively
  On maximal Valsalva maneuver: Proximal urethral rotation (degree), retrovesical angle (degree)

CONTACTS AND LOCATIONS:
Overall Officials: Murat Yassa, MD, Principal Investigator — Bartin State Hospital
Locations (1):
- Bartin State Hospital, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dogan O, Kaya AE, Pulatoglu C, Basbug A, Yassa M. A randomized comparison of a single-incision needleless (Contasure-needleless(R)) mini-sling versus an inside-out transobturator (Contasure-KIM(R)) mid-urethral sling in women with stress urinary incontinence: 24-month follow-up results. Int Urogynecol J. 2018 Sep;29(9):1387-1395. doi: 10.1007/s00192-018-3624-4. Epub 2018 Mar 16. PMID 29549394